CLINICAL TRIAL: NCT00868946
Title: A Phase 2 Treatment Protocol of Intravenous Ribavirin in Adult Subjects With Hemorrhagic Fever With Renal Syndrome (HFRS) in Landstuhl Regional Medical Center (Landstuhl, Germany) IND 16,666
Brief Title: Ribavirin for Hemorrhagic Fever With Renal Syndrome in Germany
Acronym: HFRS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-15314; BAMC HUC C.2008.197 (Other: IRB); USAMRIID HUC FY05-18 (Other: IRB)
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Hemorrhagic Fever With Renal Syndrome
Keywords: Ribavirin; Hemorrhagic Fever with Renal Syndrome; Dobrava Virus; Puumala Virus
MeSH Terms: conditions — Hemorrhagic Fever with Renal Syndrome | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment with IND Ribavirin (Experimental): All consented subjects who meet all inclusion and no exclusion criteria will enter this open label protocol and be treated with IND Virazole (Ribavirin) for 7 days with multiple dosing regime based on weight and dosage day.
  Interventions: Drug: Virazole (Ribavirin)

INTERVENTIONS:
Drug: Virazole (Ribavirin) — Duration of Subject Participation:7-day course of treatment with follow-up 28 - 60 days after first dose of IV ribavirin Route of Administration and Regimen:The drug is administered IV in a volume of 50-100 mL of normal saline to be infused over 30-40 minutes.
  Ribavirin Loading dose, 33 mg/kg (maximum dose: 2.64 g), followed by a dose of 16 mg/kg (maximum dose: 1.28 g) every 6 hours for the first 4 days (15 doses), and 8 mg/kg (maximum dose: 0.64 g) every 8 hours for the subsequent 3 days (9 doses).
  Other Names: Ribavirin

SUMMARY:
This is a treatment protocol using IND Ribavirin-there is no control group. Hemorrhagic Fever with Renal Syndrome (HFRS) is caused by a virus acquired by contact with chronically infected rodent hosts. HFRS is present throughout Europe and caused mainly by Puumala and Dobrava viruses. Treatment consists mainly of supportive care with careful attention to control of blood pressure and fluid balance and/or dialysis. Early initiation of IND Intravenous Ribavirin has been shown to be an effective treatment for HFRS and may prevent the need for dialysis. It is important to initiate therapy based on a diagnosis consistent with HFRS (determination if the disease is caused by Puumala or Dobrava virus is helpful) and a history that makes exposure likely. This study will monitor the clinical events that occur with HFRS as well as the safety and efficacy of Ribavirin.

DETAILED DESCRIPTION:
This is a Phase 2, open label study of the safety of IV Ribavirin treatment in individuals with HFRS admitted to the Landstuhl Regional Medical Center, Germany. The study will also monitor the morbidity and mortality of subjects with HFRS who are treated with IV Ribavirin. The study population will include all subjects with a probable or suspected clinical diagnosis of HFRS and meet entry criteria with a 7 day course of IV Ribavirin and a 28-60 day follow up period after the first dose of Ribavirin. In addition to treatment with Ribavirin, all subjects will be given standard supportive and symptomatic care as determined by the clinical judgment of the Principal Investigator, attending physicians or consultants who manage the subject's care at LRMC. Up to 50 subjects could potentially be enrolled in a five year time period with an expected accrual of 0-5 subjects per year. Specific inclusion/exclusion/relative exclusion criteria are a part of the protocol. Safety procedures required during 7 days of treatment include continuous cardiac monitoring, daily lab work, physical exams and vital signs.

Hemorrhagic fever with renal syndrome (HFRS) is caused by viruses in the genus Hantavirus of the family Bunyaviridae. There are four known Hantaviruses that cause HFRS: Hantaan, Seoul, Puumala, and Dobrava viruses. Hantaan virus is a spherical, enveloped virus and has been designated the prototype for the Hantavirus genus family Bunyaviridae (Schmaljohn, 1983). Serologic, morphologic, and biochemical studies have established that this virus is related to Puumala virus, Seoul virus, and other Hantaviruses (Schmaljohn, 1985). HFRS is acquired by contact with chronically infected rodent hosts, most commonly from inhalation of infected rodent excreta (urine, saliva, and feces) but also reported from rodent bites. In Europe, HFRS is caused mainly by Puumala and Dobrava viruses, with Puumala virus responsible for most cases. Puumala virus, the cause of nephropathia epidemica (NE) in Scandinavia (also France, Germany, Belgium, Scotland, and Italy), is transmitted by Clethrionomys glareolus (mole) [HFRS manual Niklasson]. HFRS from Puumala virus is associated with a mortality rate of <0.5%. Oliguria is reported in 40% of cases, and severe renal insufficiency is generally observed in 3 to 9% cases [HFRS manual Lahdevirta]. However, a report from HFRS due to Puumala virus in Germany was associated with severe renal disease necessitating dialysis in 4/15 (26% cases) [Rasche et al, 2004)].

Dobrava virus, the cause of a severe form of HFRS mainly in the Balkan Peninsula (Hungary, Bulgaria, Albania, the former Yugoslavia, and Greece) but also in Russia in areas west of the Ural Mountains, is transmitted by the rodent host Apodemus flavicollis (yellow-necked field mouse), and associated with a mortality rate of 5%-35% {HFRS manual Tatjana; HFRS manual Tkachenko]. Less data is available on Dobrava virus, but the morbidity and mortality is expected to be similar to HFRS caused by Hantaan virus, or perhaps more severe. In one study of HFRS in Greece felt to be secondary to Dobrava virus, 37% cases required dialysis and 15% cases resulted in death (Antoniadis et al, 1989).

Disease from Dobrava virus has a similar severity and presentation as disease from Hantaan virus. However, HFRS from Puumala has a lower death rate and dialysis rate and the risk of IV Ribavirin in treatment for HFRS, in particular, must be measured against the benefit of treatment. The decision to start IND IV Ribavirin will be based on whether the HFRS is likely to be Dobrava virus versus Puumala virus based on epidemiological data of past or ongoing outbreaks of HFRS in that geographical area. Observation with supportive care without the use of IND IV Ribavirin is the generally recommended medical management of HFRS from Puumala virus due to the lower morbidity and mortality associated with HFRS from Puumala virus.

While most cases in HFRS in Europe will be from Puumala and Dobrava viruses, the experience with IV ribavirin has been mainly with HFRS caused by Hantaan and Seoul viruses in Southeast Asia. All hantaviruses have in vitro sensitivity to IV ribavirin. The data for IV ribavirin for HFRS caused by hantaviruses in Europe is based on the experience with HFRS from Hantaan and Seoul viruses.

Ribavirin is licensed in the United States in aerosol form for the treatment of severe lower respiratory tract infection in children and in the oral formulation in combination with recombinant interferon alpha for the treatment of chronic hepatitis C infection. The intravenous formulation of ribavirin is not licensed in the U.S. IV Ribavirin for the treatment of HFRS is used under IND 16,666.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the case definition for a probable or suspected case.
2. Has read and signed the Informed Consent.
3. Is at least 18 years of age (17, if active military) and not greater than 65 years of age.
4. Has a blood sample drawn and a type and cross-match ordered for transfusion.
5. Agrees to collection of required specimens.
6. Agrees to report any Adverse Event, Serious and Unexpected Adverse Events which may or may not be associated with administration of the drug for the duration of the study.
7. Agrees to a follow-up visit and to donate blood and urine specimens at day 10, day 14 and between days 28 and 60 after their first dose of IV Ribavirin and to all follow-up visits for anemia or other medical conditions as required by the attending physician.
8. Woman of childbearing age has a negative pregnancy test and agrees not to become pregnant during treatment and for 7 months after receiving Ribavirin. Treatment will be a maximum of 25 doses given over a one week time period. At least two reliable forms of effective contraception, including one barrier method, must be utilized during treatment and during the 7 months post-treatment period.
9. Man agrees not to have intercourse with a pregnant woman during treatment and for 7 months after receiving Ribavirin, and take precautions to avoid producing pregnancies in female partners during and for 7 months after receiving Ribavirin.

   Treatment will be a maximum of 25 doses given over a one week time period. At least two reliable forms of effective contraception, including one barrier method, must be utilized during the treatment and during the 7 month post-treatment period.
10. Has a hemoglobin of 10 g/dL or higher before starting IV Ribavirin.

Exclusion Criteria:

1. Has know intolerance to Ribavirin
2. Is pregnant
3. Is irreversibly ill on presentation, as defined by presence of profound shock (shock which does not respond to supportive therapy within 3 hours after admission).
4. Has history of hemoglobinopathies (i.e., sickle-cell anemia or thalassemia major)
5. Has history of autoimmune hepatitis
6. Has a calculated serum creatinine clearance of < 20 mL/min
7. Has hemoglobin less than 10 g/dL that cannot be corrected to 10 g/dL before initiation of IV Ribavirin.
8. Is considered as New York Heart Association Cardiac functional capacity of Class II or greater for ASHD and CHF.
9. Has known cardiac conduction defects that may predispose to arrhythmias such as Wolfe-Parkinson-White Syndrome (WPW); or a history of bradyarrhythmias such as sick sinus syndrome or second degree heart block and no pacemaker.
10. Has sinus bradycardia of less than 40 beats per minute (or sinus bradycardia less than 50 beats per minute if the individual is not known to have a low resting heart rate related to physical conditioning). If an individual develops heart rate of less than 35 beats per minute while on IV Ribavirin, the IV Ribavirin may be discontinued by the physician.
11. Is currently being treated with Didanosine (ddI). DdI must be discontinued before starting IV Ribavirin.

Relative exclusion criteria:

1. History of gout or tophaceous gout
2. Use of drugs known to result in bradyarrhythmias (certain betablockers and calcium channel blockers)
3. Creatinine clearance of 20 to 30 mL/min

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of subject who develop oliguria | 5 years
  Number of subject who develop oliguria (≤ 400 mL of urine in a 24-hour period), who require hemodialysis, who have cardiac arrhythmias, or who experience severe hemorrhage [results in hypotension (< 90 mm Hg systolic blood pressure) or hemorrhagic shock]. Subject mortality will be evaluated.
Number of mortalities | 5 years

SECONDARY OUTCOMES:
Number and type of adverse events for all subjects. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Rini, Principal Investigator — Landstuhl Regional Medical Center
Locations (1):
- Landstuhl Regional Medical Center, Landstuhl, APO AE, Germany